CLINICAL TRIAL: NCT04504864
Title: Low-dose Aspirin Therapy in Patients With Non-Cardioembolic Ischemic Stroke and Microbleeds
Brief Title: Low-dose Aspirin Therapy in Patients With Ischemic Stroke and Microbleeds
Acronym: AIM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Shaanxi Provincial People's Hospital (Other); The First Affiliated Hospital of Jiaotong University (Unknown); Tang-Du Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xi'an Central Hospital (Other); Xiangyang Central Hospital (Other); Baoji Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY20202059-F-1
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; microbleeds; Clinical trial; Aspirin
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose aspirin (Experimental): Management policy is to use 50 mg aspirin per day as a secondary prevention strategy for patients with non-cardioembolic ischemic stroke and microbleeds. 50mg aspirin is recommended by the guideline of ASA/AHA in prevention of stroke. But this dose is rarely used clinically, especially in East Asia area.
  Interventions: Drug: low-dose aspirin
- conventional-does aspirin (Active Comparator): Management policy is to use 100 mg aspirin per day as a secondary prevention strategy for patients with non-cardioembolic ischemic stroke and microbleeds. 100mg aspirin is recommended by the guideline of ASA/AHA in prevention of stroke, and this dose is widely used clinically.
  Interventions: Drug: conventional-does aspirin

INTERVENTIONS:
Drug: low-dose aspirin — 50mg aspirin is used to prevent recurrent stroke.
  Arms: low-dose aspirin
Drug: conventional-does aspirin — 100mg aspirin is used to prevent recurrent stroke.
  Arms: conventional-does aspirin

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of low-dose (50mg) aspirin as a secondary prevention drug in patients with Non-Cardioembolic Ischemic Stroke accompanied by cerebral microbleeds.

DETAILED DESCRIPTION:
Cerebral microbleeds are caused by microvascular lesions in the brain, which is a subclinical deposition of hemosiderin after the damage of microvascular. Aspirin is the most widely used anti-thrombotic drug in the secondary prevention of patients with non-cardioembolic ischemic stroke. Studies have shown that conventional doses of aspirin can increase the incidence of intracranial hemorrhage in ischemic stroke patients with cerebral microbleeds. For such patients, how to carry out effective and safe anti-thrombotic therapy is still unclear.

The AIM study aims to provide reliable data on the effects of low-dose Aspirin (50mg target recruitment 200) in patients with non-cardioembolic ischemic stroke and cerebral microbleeds compared to conventional dose (100mg target recruitment 200). Patients presenting with acute (<3 weeks) non-cardioembolic ischemic stroke and microbleeds (≧1 microbleeds in SWI scans) will be randomly assigned to the secondary stroke prevention therapy of low-dose or conventional dose aspirin for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cerebral infarction diagnosed clinically as non-cardioembolic ischemic stroke;
2. Age ≥ 18 years;
3. Onset time ≤ 3 weeks;
4. At least one cerebral microbleeds lesion was found on SWI;
5. Informed consent was signed.

Exclusion Criteria:

1. Patients with symptomatic intracranial hemorrhage;
2. No microbleeds or bleeding lesion > 10 mm was found on SWI;
3. Vascular malformations, tumors, abscesses or other major non ischemic brain diseases were present;
4. Clear anticoagulant indications (such as atrial fibrillation);
5. There are contraindications for aspirin use;
6. The focus of microbleeds is limited to the cortex or other evidence suggests that the patient has cerebral amyloid angiopathy;
7. Patients with coronary heart disease or other diseases need to take antiplatelet drugs;
8. Serious systemic diseases;
9. Refusal to sign informed consent or poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Increase of cerebral microbleeds | 6 months after onset
  How many cerebral microbleeds increased after 6 months of aspirin treatment. Cerebral microbleeds will be detected by MR-SWI in the acute stage and 6 months after the onset of stroke.

SECONDARY OUTCOMES:
Stroke recurrence rate | 6 months after onset
  recurrence rate of ischemic stroke
The incidence of cerebral hemorrhage | 6 months after onset

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jiang, Ph.D, Study Director — Department of Neurology, Xijing Hospital, Fourth Military Medical University
Locations (6):
- China (6):
  - Baoji Central Hospital, Baoji, Shaanxi
  - Department of Neurology, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi'an, Shaanxi
  - Xi'an Central Hospital, Xi'an, Shaanxi
  - Xianyang Central Hospital, Xianyang, Shaanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Background] Shoamanesh A, Pearce LA, Bazan C, Catanese L, McClure LA, Sharma M, Marti-Fabregas J, Anderson DC, Kase CS, Hart RG, Benavente OR; SPS3 Trial Investigators. Microbleeds in the Secondary Prevention of Small Subcortical Strokes Trial: Stroke, mortality, and treatment interactions. Ann Neurol. 2017 Aug;82(2):196-207. doi: 10.1002/ana.24988. Epub 2017 Jul 19. PMID 28681535
- [Background] Kleinig TJ. Associations and implications of cerebral microbleeds. J Clin Neurosci. 2013 Jul;20(7):919-27. doi: 10.1016/j.jocn.2012.12.002. Epub 2013 May 24. PMID 23707603
- [Background] Wilson D, Charidimou A, Ambler G, Fox ZV, Gregoire S, Rayson P, Imaizumi T, Fluri F, Naka H, Horstmann S, Veltkamp R, Rothwell PM, Kwa VI, Thijs V, Lee YS, Kim YD, Huang Y, Wong KS, Jager HR, Werring DJ. Recurrent stroke risk and cerebral microbleed burden in ischemic stroke and TIA: A meta-analysis. Neurology. 2016 Oct 4;87(14):1501-1510. doi: 10.1212/WNL.0000000000003183. Epub 2016 Sep 2. PMID 27590288
- [Background] Benedictus MR, Prins ND, Goos JD, Scheltens P, Barkhof F, van der Flier WM. Microbleeds, Mortality, and Stroke in Alzheimer Disease: The MISTRAL Study. JAMA Neurol. 2015 May;72(5):539-45. doi: 10.1001/jamaneurol.2015.14. PMID 25798556
- [Background] Akhtar N, Salam A, Kamran S, D'Souza A, Imam Y, Bermejo PG, Wadiwala MF, Own A, ElSotouhy A, Vattoth S, Bourke P, Bhutta Z, Joseph S, Santos M, Khan RA, Shuaib A. Pre-existing Small Vessel Disease in Patients with Acute Stroke from the Middle East, Southeast Asia, and Philippines. Transl Stroke Res. 2018 Jun;9(3):274-282. doi: 10.1007/s12975-017-0578-7. Epub 2017 Nov 3. PMID 29101611
- [Background] Charidimou A, Shams S, Romero JR, Ding J, Veltkamp R, Horstmann S, Eiriksdottir G, van Buchem MA, Gudnason V, Himali JJ, Gurol ME, Viswanathan A, Imaizumi T, Vernooij MW, Seshadri S, Greenberg SM, Benavente OR, Launer LJ, Shoamanesh A; International META-MICROBLEEDS Initiative. Clinical significance of cerebral microbleeds on MRI: A comprehensive meta-analysis of risk of intracerebral hemorrhage, ischemic stroke, mortality, and dementia in cohort studies (v1). Int J Stroke. 2018 Jul;13(5):454-468. doi: 10.1177/1747493017751931. Epub 2018 Jan 17. PMID 29338604
- [Background] Charidimou A, Imaizumi T, Moulin S, Biffi A, Samarasekera N, Yakushiji Y, Peeters A, Vandermeeren Y, Laloux P, Baron JC, Hernandez-Guillamon M, Montaner J, Casolla B, Gregoire SM, Kang DW, Kim JS, Naka H, Smith EE, Viswanathan A, Jager HR, Al-Shahi Salman R, Greenberg SM, Cordonnier C, Werring DJ. Brain hemorrhage recurrence, small vessel disease type, and cerebral microbleeds: A meta-analysis. Neurology. 2017 Aug 22;89(8):820-829. doi: 10.1212/WNL.0000000000004259. Epub 2017 Jul 26. PMID 28747441
- [Background] Werring DJ, Charidimou A; authors. Response by Werring and Charidimou to Letter Regarding Article, "Microbleeds, Cerebral Hemorrhage, and Functional Outcome After Stroke Thrombolysis: Individual Patient Data Meta-Analysis". Stroke. 2017 Nov;48(11):e332. doi: 10.1161/STROKEAHA.117.019038. Epub 2017 Oct 13. No abstract available. PMID 29030477
- [Background] Kim BJ, Kwon SU, Park JH, Kim YJ, Hong KS, Wong LKS, Yu S, Hwang YH, Lee JS, Lee J, Rha JH, Heo SH, Ahn SH, Seo WK, Park JM, Lee JH, Kwon JH, Sohn SI, Jung JM, Navarro JC, Kim HY, Kim EG, Kim S, Cha JK, Park MS, Nam HS, Kang DW; PICASSO Investigators. Cilostazol Versus Aspirin in Ischemic Stroke Patients With High-Risk Cerebral Hemorrhage: Subgroup Analysis of the PICASSO Trial. Stroke. 2020 Mar;51(3):931-937. doi: 10.1161/STROKEAHA.119.023855. Epub 2019 Dec 20. PMID 31856691
- [Background] Poels MM, Ikram MA, van der Lugt A, Hofman A, Krestin GP, Breteler MM, Vernooij MW. Incidence of cerebral microbleeds in the general population: the Rotterdam Scan Study. Stroke. 2011 Mar;42(3):656-61. doi: 10.1161/STROKEAHA.110.607184. Epub 2011 Feb 9. PMID 21307170
- [Result] Lau KK, Wong YK, Teo KC, Chang RSK, Tse MY, Hoi CP, Chan CY, Chan OL, Cheung RHK, Wong EKM, Kwan JSK, Hui ES, Mak HKF. Long-Term Prognostic Implications of Cerebral Microbleeds in Chinese Patients With Ischemic Stroke. J Am Heart Assoc. 2017 Dec 7;6(12):e007360. doi: 10.1161/JAHA.117.007360. PMID 29217662
- [Result] Jia C, Wei C, Hu M, Xu J, Niu K, Zhang C, Lv P, Li L, Dong Y. Correlation between antiplatelet therapy in secondary prevention of acute cerebral infarction and cerebral microbleeds: A susceptibility-weighted imaging (SWI) study. J Xray Sci Technol. 2018;26(4):623-633. doi: 10.3233/XST-17361. PMID 29562586
- [Result] Lau KK, Lovelock CE, Li L, Simoni M, Gutnikov S, Kuker W, Mak HKF, Rothwell PM. Antiplatelet Treatment After Transient Ischemic Attack and Ischemic Stroke in Patients With Cerebral Microbleeds in 2 Large Cohorts and an Updated Systematic Review. Stroke. 2018 Jun;49(6):1434-1442. doi: 10.1161/STROKEAHA.117.020104. Epub 2018 May 10. PMID 29748422